CLINICAL TRIAL: NCT03898791
Title: Phase 1b Study of LY3295668 Erbumine Monotherapy in Patients With Platinum-Sensitive, Extensive-Stage Small-Cell Lung Cancer
Brief Title: A Study of LY3295668 Erbumine in Participants With Extensive-stage Small-Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17248; J1O-MC-JZHB (Other: Eli Lilly and Company); 2018-003485-14 (EudraCT Number)
Record Dates: First submitted 2019-04-01; First posted 2019-04-02 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Small Cell Lung Cancer
Keywords: aurora kinase A; kinase; aurora A; aurora kinase inhibitor; aurora kinase A inhibitor; kinase inhibitor; AURKA; AurA
MeSH Terms: conditions — Small Cell Lung Carcinoma; Epilepsy | interventions — LY3295668 erbumine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3295668 Erbumine Cohort A (Experimental): LY3295668 erbumine administered orally.
  Interventions: Drug: LY3295668 Erbumine
- LY3295668 Erbumine Cohort B (Experimental): LY3295668 erbumine administered orally.
  Interventions: Drug: LY3295668 Erbumine
- LY3295668 Part JP (Experimental): LY3295668 erbumine administered orally.
  Interventions: Drug: LY3295668 Erbumine

INTERVENTIONS:
Drug: LY3295668 Erbumine — oral capsules

SUMMARY:
The purpose of this study is to determine the recommended phase 2 dose of LY3295668 erbumine in participants with platinum-sensitive, extensive-stage small-cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological evidence of a diagnosis of platinum sensitive small cell lung cancer that is extensive stage.
* Have adequate organ function.
* Have a performance status (PS) of ≤1 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Have discontinued previous treatments for cancer.
* Are able to swallow capsules.

Exclusion Criteria:

* Currently enrolled in a clinical study.
* Have a serious concomitant systemic disorder.
* Have a symptomatic human immunodeficiency virus infection or symptomatic activated/reactivated hepatitis B or C.
* Have a significant cardiac condition.
* Have previously received an aurora kinase inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose Reductions | Baseline through Cycle 1 (28 Day Cycle)
  Number of Participants with Dose Reductions
Objective Response Rate (ORR): Percentage of Participants Who Achieve Complete Response (CR) or Partial Response (PR) | Baseline through Measured Progressive Disease (Estimated up to 20 Months)
  ORR: Percentage of participants who achieve CR or PR
Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of LY3295668 Erbumine | Predose Cyce 1 Day 1 through Cycle 2 Day 1 (28 Day Cycles)
  PK: AUC of LY3295668 Erbumine
Duration of Response (DoR) | Date of CR or PR to Date of Disease Progression or Death Due to Any Cause (Estimated up to 20 Months)
  DoR

SECONDARY OUTCOMES:
PK: Maximum Concentration (Cmax) of LY3295668 Erbumine | Predose Cyce 1 Day 1 through Cycle 2 Day 1 (28 Day Cycles)
  PK: Cmax of LY3295668 Erbumine
Best Overall Response (BOR): Percentage of Participants with CR, PR, Stable Disease (SD), or Progressive Disease (PD) | Baseline to Date of Objective Disease Progression (Estimated up to 20 Months)
  BOR
Disease Control Rate (DCR): Percentage of Participants with a Best Overall Response of CR, PR, and SD | Baseline through Measured Progressive Disease (Estimated up to 20 Months)
  DCR

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (40):
- United States (16):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Rocky Mountain Cancer Center, Denver, Colorado
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University Medical School, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute- Carolinas Medical Center, Charlotte, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute, Greenville, South Carolina
  - Texas Oncology Cancer Center, Austin, Texas
  - Texas Oncology Fort Worth, Fort Worth, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - US Oncology, The Woodlands, Texas
  - Tyler Cancer Center, Tyler, Texas
- Belgium (4):
  - Grand Hopital de Charleroi-Site Notre-Dame, Charleroi
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
  - AZ Delta, Roeselare
- France (6):
  - Institut Bergonie, Bordeaux
  - Centre Georges Francois Leclerc, Dijon
  - Centre de Lutte Contre le Cancer Leon Berard, Lyon
  - APHM Hôpital de la Timone, Marseille
  - Institut Curie, Paris
  - Institut de Cancérologie de l'Ouest Centre René Gauducheau, Saint-Herblain
- National Cancer Center Hospital, Chuo-Ku, Tokyo, Japan
- South Korea (3):
  - Severance Hospital Yonsei University Health System, Seoul, Korea
  - Samsung Medical Center, Seoul, Korea
  - Asan Medical Center, Seoul
- Spain (6):
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga, Andalusia
  - Institut Catala d'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Fe de Valencia, Valencia
- Turkey (Türkiye) (2):
  - Dr.Abdurrahman Yurtaslan Ankara Oncology Training & Res Hosp, Ankara
  - Ege University Faculty of Medicine, Izmir
- United Kingdom (2):
  - Guys/St. Thomas Hospital, London, Surrey
  - Royal Marsden Hospital, Sutton, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of LY3295668 Erbumine in Participants With Extensive-stage Small-Cell Lung Cancer — https://trials.lillytrialguide.com/en-US/trial/466NNvH4TeYW4gBJz8K9Xp